CLINICAL TRIAL: NCT02591797
Title: Effectiveness of Hand/Eyes/Mouth Behavior Management Technique in Anxiety, Pain and Behavior Levels During an Inferior Alveolar and Lingual Nerve Block Procedure in Preschool Children: a Randomized Clinical Trial
Brief Title: Effectiveness of Hand/Eyes/Mouth Behavior Management Technique During Local Anesthesia in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Ana María Leyda Menéndez, Dr. Associate Professor to the Pediatric Dentistry Master, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMLUCHBR
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Dental Anxiety; Pain; Infant Behavior; Heart Rate and Rhythm Disorders
Keywords: pain; Infant Behavior; Heart rate; Dental Anxiety
MeSH Terms: conditions — Pain; Infant Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- "hand-eye-mouth" technique (Experimental): "hand-eye-mouth" (MOB) seeks to focus the patient in performing a sequence of movements in a fun way so that your attention is diverted from the puncture dental needle, also it seeks to the patient does not see the needle. The operator prior to infiltrate local anesthetic teaches the child a "game" to put "the sleepy little water".After explain a first time, the sequence once or twice is repeated until the patient has mastered. We call this test. When we apply the anesthetic, the entire sequence must be repeated as in trials with the same tranquility and in the same tone of the game. The operator will use this technique during the inferior alveolar and lingual nerve block procedure
  Interventions: Procedure: inferior alveolar and lingual nerve block procedure
- Conventional technique (Active Comparator): the operator will explain how he/she will do the inferior alveolar and lingual nerve block procedure in phrases appropriates to the child. Then quietly cover the child´s field of view by hand during the inferior alveolar and lingual nerve block
  Interventions: Procedure: inferior alveolar and lingual nerve block procedure

INTERVENTIONS:
Procedure: inferior alveolar and lingual nerve block procedure — The needle is inserted laterally to the pterygomandibular pit at its deepest point without noticing any resistance. In children the positioning of the syringe must be perpendicular, between the canine and the first molar on the opposite side and puncture is performed slightly below the occlusal plane. It was initially deposited 2/3 anesthetic carpule solution and then the needle is slightly recede depositing there the remaining third of anesthetic solution.
  The application of anesthesia shall be in accordance with the following guidelines:
  1. Topical Anesthetic: Benzocaine 20% (Hurricaine, Clarben Laboratories SA, Madrid, Spain).
  2. Dental Needle: short needles (21mm/30g) (Octoplus, Clarben Laboratories SA, Madrid, Spain)
  3. anesthetic: lidocaine hydrochloride 2% with epinephrine 1: 100,000 (2% XILOCAINE, Dentsply, Spain).
  4. Syringe: carpule syringe-conventional harpoon with suction system.
  Other Names: inferior alveolar and lingual nerve block

SUMMARY:
This will be a randomized, controlled, parallel-group clinical trial. The aim of this studio will be to evaluate the effectiveness of "Hands/Eyes/mouth" behavior management technique versus a conventional technique (covering the patient´s vision) during an inferior alveolar and lingual nerve block in preschool children referred for treatment at the School of Dentistry, Cardenal Herrera CEU University (Valencia, Spain). The sample will consist of 52 children from 3 years old to 5 years 11 months old who need dental pulp treatment and/or tooth extraction of primary molars. Preschool children with no history of allergies to Lidocaine or systemic/neurological diseases and who did not take local anesthesia before the study will be include in this research.

DETAILED DESCRIPTION:
Children will be randomly allocated to treatment groups (n=26 for each group) according to the technique: 1)"Hands/Eyes/mouth" and 2) Conventional. Anxiety and pain will be evaluated by the Scale of facial Image (EIF) and Wong-Baker Pain Scale, respectively. The cooperation of the patient will be evaluated by behavioral Scale Frank

ELIGIBILITY:
Inclusion Criteria:

* Preschool children with severe dental caries who need dental pulp treatment and/or tooth extraction of inferior primary molars

Exclusion Criteria:

* Preschool children with history of allergies to lidocaine (local anesthetic)
* Preschool children with systemic or neurological diseases
* Preschool children who have received local dental anesthesia before this study
* Preschool children who do not understand Spanish or Valencian language

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Preschool children´s anxiety levels-Facial Image Scale (FIS) | Baseline
  The children will be asked to point at which face they felt most like at that moment (row of five faces ranging from very happy to very unhappy-FIS)

SECONDARY OUTCOMES:
Preschool children´s pain levels-Wong Baker Faces Pain Scale | At the end of local anesthesia procedure (2 minutes)
  The children will be asked to point at which face they felt most like at that moment (row of six faces ranging from very happy-does not hurt to very unhappy-hurt as much as you can imagine)

OTHER OUTCOMES:
Preschool children´s behavior-Frank behavioral rating Scale | baseline and during the local anesthesia procedure (2 minutes)
  It will be evaluated children´s behavior (definitely negative, negative,definitely positive, positive)during the local anethesia procedure
Heart rates | baseline and during the local anesthesia procedure (2 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ribelles Llop, PhD, Study Director — Director of Pediatric Dentistry Master. Cardenal Herrera CEU University
Locations (1):
- Facultad de Odontología. Universidad Cardenal Herrera CEU, Valencia, Spain

REFERENCES:
- [Derived] Leyda-Menendez AM, Vidigal EA, Abanto J, Ribelles-Llop M. Efficacy of two behavioural management techniques during inferior alveolar nerve block administration in pre-school children: a randomised clinical trial. Eur Arch Paediatr Dent. 2023 Feb;24(1):85-93. doi: 10.1007/s40368-022-00758-y. Epub 2022 Oct 19. PMID 36260279